CLINICAL TRIAL: NCT00879775
Title: Efficacy of Caffeine as an Adjuvant to Opioid Therapy in Cancer Pain: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of Caffeine Injection as an Adjuvant to Opioid Therapy in Cancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Research Foundation (Other)
Collaborators: Korea University Guro Hospital (Other)
Responsible Party: Sang-Yeon Suh, Dongguk University Ilsan Hospitial
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: E00058; GR0857-006 (Other: Korea University Guro Hospital); SuYeon2009-08 (Other: National Health Insurance Corporation Ilsan Hospital)
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2009-09

CONDITIONS: Cancer; Pain
Keywords: Pain; Cancer patients; Caffeine; Adjuvant analgesics; Sedation; Confusion; Quality of life; Fatigue
MeSH Terms: conditions — Neoplasms; Pain; Confusion; Fatigue | interventions — Caffeine; caffeine, sodium benzoate drug combination; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Experimental): Intravenous injections of 200mg of caffeine with 100ml of normal saline over 1 hour
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Intravenous injections of 100ml of normal saline over 1 hour
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Caffeine — Intravenous injection of caffeine 200mg with 100ml of normal saline over 1 hour, once a day, for two days.
  Other Names: Caffeine sodium benzoate
  Arms: Caffeine
Drug: Normal saline — Intravenous injections of 100ml of normal saline over 1 hour, once a day, for two days
  Other Names: 0.9% saline
  Arms: Placebo

SUMMARY:
Pain is a most common symptom and it has a high impact on quality of life in cancer patients. Many cancer patients have received opioid therapy, but also many of them have suffered from side effects of opioids. Drowsiness and confusion are common side effects of opioids. Caffeine is a well known psychostimulant,and it is widely used as an analgesics. Thus, the investigators aimed to prove the efficacy of intravenous caffeine administration as an adjuvant analgesics to opioids. At the same time, the investigators tried to find that the side effects of opioids could be ameliorated by caffeine.

DETAILED DESCRIPTION:
Previous studies on cancer pain lacked assessment of quality of life. And most of previous studies on cancer pain did not give attention to symptoms accompanied with pain. We include such variables as outcome measures, and aimed to evaluate the efficacy and the safety of intravenous caffeine in advanced cancer inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (Stage IV) cancer inpatients
* Adults aged over 18 years
* Patients who have received opioid therapy and whose pain scales are under 6 (by numeric rating scale)
* Patients who do not take caffeine beverage 48 hours before study period
* Volunteers who provided written informed consent

Exclusion Criteria:

* Sensitivity (palpitation,headache,irritability,insomnia) to caffeine
* Uncontrolled hypertension and/or heart disease
* Liver failure (alanine aminotransferase >= 100 IU/L)
* Kidney failure (serum creatinine >= 2.0 mg/dL)
* Patients taken theophylline
* Gastroesophageal reflux disease
* Chronic glaucoma
* Cognitive impairment
* Progressive pain over 7 (by numeric rating scale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Yeon Suh, M.D.,Ph.D, Principal Investigator — DongGuk University
Locations (2):
- South Korea (2):
  - National Health Insurance Corporation Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Korea University Guro Hospital, Seoul

REFERENCES:
- [Background] Mercadante S, Serretta R, Casuccio A. Effects of caffeine as an adjuvant to morphine in advanced cancer patients. A randomized, double-blind, placebo-controlled, crossover study. J Pain Symptom Manage. 2001 May;21(5):369-72. doi: 10.1016/s0885-3924(01)00249-4. PMID 11369156
- [Background] Manfredi PL, Gonzales GR. Symptomatic uses of caffeine in patients with cancer. J Palliat Care. 2003 Spring;19(1):63-5. No abstract available. PMID 12710118
- [Background] Bruera E, Watanabe S. Psychostimulants as adjuvant analgesics. J Pain Symptom Manage. 1994 Aug;9(6):412-5. doi: 10.1016/0885-3924(94)90179-1. PMID 7963794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 participants were screened. 1 did not meet criteria.
Period: Overall Study
Arm/Group | Caffeine | Placebo
Started | 20 | 21
Completed | 18 | 20
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 63.40 (11.76) | 67.83 (9.76) | 65.67 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20 | 21 | 41
Symptom score [Mean (Standard Deviation); unit: scores] — Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; a higher score represents a higher level of symptoms.
  scores
    Pain | 3.25 (1.06) | 3.52 (1.12) | 3.39 (1.09)
    Drowsiness | 4.05 (1.57) | 4.24 (1.54) | 4.15 (1.54)
    Nausea | 2.20 (1.19) | 2.33 (1.23) | 2.27 (1.21)
    Sleep | 4.20 (1.96) | 3.90 (1.86) | 4.05 (1.90)
    Sadness | 4.55 (1.39) | 4.23 (1.51) | 4.39 (1.45)
    Fatigue | 4.50 (1.60) | 4.47 (1.56) | 4.49 (1.57)
    Confusion | 1.95 (1.57) | 2.52 (1.50) | 2.24 (1.55)
Health-related quality of life [Mean (Standard Deviation); unit: scores] — Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; a higher score represents a better health-related quality of life.
  scores | 4.30 (1.34) | 4.19 (1.12) | 4.24 (1.22)
Impact of symptom burden to daily life (by MD Anderson Symptom Inventory-Korean) [Mean (Standard Deviation); unit: scores] — Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; a higher score represents a higher level of impact of symptom burden to daily life.
  scores
    Daily living | 5.00 (2.12) | 5.90 (1.86) | 5.46 (2.03)
    Mode | 5.90 (1.51) | 6.09 (1.33) | 6.00 (1.41)
    Work | 6.25 (2.14) | 6.90 (1.64) | 6.59 (1.91)
    Interpersonal relationship | 4.80 (2.01) | 5.09 (1.54) | 4.95 (1.77)
    Gait ability | 4.45 (2.50) | 5.61 (1.93) | 5.05 (2.28)
    Life enjoyment | 6.70 (1.97) | 7.66 (1.55) | 7.20 (1.82)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating of Scale (From 0 to 10) of Pain and Possible Side Effects (Drowsiness, Confusion, Nausea) of Opioids
Description: Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; higher scores represent higher levels of pain, and possible side effects (drowsiness, confusion, nausea) of opioids.
Time Frame: two days
Population: intention to treat
Measure: Mean (Standard Deviation); unit: scores
Units Other Than Participants: Symptoms
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 20 | 21
Number analyzed (Symptoms) | 18 | 20
scores
  Pain | 2.22 (1.22) | 3.10 (1.17)
  Drowsiness | 2.83 (1.92) | 3.05 (1.57)
  Confusion | 1.89 (1.68) | 2.20 (1.36)
  Nausea | 2.28 (1.41) | 1.80 (0.77)

2. Secondary Outcome: Degree of Fatigue at the Point of Time With Numeric Rating Scale From 0 to 10
Description: Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; a higher score represents a higher level of fatigue.
Time Frame: two days
Population: intention to treat
Measure: Mean (Standard Deviation); unit: scores
Units Other Than Participants: Symptoms
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 20 | 21
Number analyzed (Symptoms) | 18 | 20
scores | 3.61 (1.88) | 3.55 (1.50)

3. Secondary Outcome: Health-related Quality of Life
Description: Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; a higher score represents a better health-related quality of life.
Time Frame: two days
Population: intention to treat
Measure: Mean (Standard Deviation); unit: scores
Units Other Than Participants: Symptoms
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 20 | 21
Number analyzed (Symptoms) | 18 | 20
scores | 4.83 (1.30) | 4.45 (0.89)

4. Secondary Outcome: Impact of Symptom Burden to Daily Life (by MD Anderson Symptom Inventory-Korean)
Description: Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; a higher score represents a higher level of impact of symptom burden to daily life.
Time Frame: two days
Population: intention to treat
Measure: Mean (Standard Deviation); unit: scores
Units Other Than Participants: Symptoms
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 20 | 21
Number analyzed (Symptoms) | 18 | 20
scores
  Daily living | 5.17 (2.07) | 5.95 (1.82)
  Mood | 5.61 (1.69) | 5.60 (1.54)
  Work | 5.56 (1.85) | 6.75 (1.55)
  Interpersonal relationship | 4.61 (1.79) | 4.65 (1.69)
  Gait ability | 4.39 (2.36) | 5.50 (2.12)

5. Primary Outcome: Numeric Rating of Scale (From 0 to 10) of Possible Sleep Disturbance of Opioids
Description: Scores were measured by Numeric Rating Scale. Scores range from 0 to 10; a higher score represents a higher level of sleep disturbance.
Time Frame: two days
Measure: Mean (Standard Deviation); unit: scores
Units Other Than Participants: Symptoms
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 20 | 21
Number analyzed (Symptoms) | 18 | 20
scores | 3.53 (1.81) | 3.80 (1.79)

ADVERSE EVENTS:
Arm/Group | Caffeine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine (N=18) | Placebo (N=20)
Blood pressure elevation (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No